CLINICAL TRIAL: NCT05022420
Title: SAfety and TOlerance of the Biopsies in Auto-immune Rare dIseases
Acronym: SATORI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: SATORI (29BRC21.0089)
Record Dates: First submitted 2021-08-25; First posted 2021-08-26 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Tolerance; Biopsy Site Itching

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Salivary gland biospy,: 100 Salivary gland biospy use for the diagnosis of sjogern disease or other auto-immune disease.
- muscular biopsy,: muscular biospy use for the diagnosis of muscular auto-immune disease.
- neuro muscular biospy: neuro muscular biospy use for the diagnosis of vasculitis,muscular auto-immune disease or neuro-muscumar auto-immune disease
- temporal arteries biospy: temporal arteries biospy uses for the diagnosis of giant cell arteritis

SUMMARY:
Biopsies are performed in several autoimmune diseases to diagnose or classify them Tolerance and information of the patients have been poorly evlauated our objective is to evaluate tolerance and information of the patients after the biopsies for salivary gland, temporal arteries and neuromuscular.

DETAILED DESCRIPTION:
patinets that benefited of arterial temporal biospy or salivary gland biospy or muscuar biopsy or neuro muscular biospy for his auto -mmune disease will be included and fill standardized questionnaires concerning tolerance, information and side effect at inclusion , day 7 and day 30 after the biopsy data will be analysed to evaluate information, tolerance and risk factor af side effect

ELIGIBILITY:
Inclusion Criteria:

* biospy required for the diagnsis or follow up aged of more than 18 non opposition form

Exclusion Criteria:

* unable to consent demencia unable to fill the form and questionnaire patient Under juridical protection refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients that underwent a biospy for his auto-immune rare disease
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2025-02-18 (Estimated); Study Completion 2025-02-18 (Estimated)

PRIMARY OUTCOMES:
tolerance of each type of biopsy | tolerance at day 7 after the biospy was performed
  tolerance based on a standardized patient 's questionnaire

SECONDARY OUTCOMES:
tolerance of each type of biopsy 30 days after | tolerance at day 30 and at inclusion after the biospy was performed
  tolerance based on a standardized patient 's questionnaire
evaluation of the qualitiy of patient's information at inclusion | questionnaire at inclusion
  standardized questionnaire at inclusion
risk factor of sied effect of each biospy | standardized questionnaire at inclusion, day 7 and 30
  standardized questionnaire

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU d'ANGERS, Angers
  - CHU de Bordeaux, Bordeaux
  - CHRU de Brest, Brest
  - CHU de LILLE, Lille
  - CHU de Marseille, Marseille
  - Hôpital de la Salpétrière, Paris
  - CH de Quimper, Quimper
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.